CLINICAL TRIAL: NCT05406505
Title: Effect of Adjuvant Dapagliflozin on Improving the Treatment of Congestion in Patients With Acute Heart Failure (DAPA-RESPONSE-AHF)
Brief Title: Effect of Dapagliflozin in Patients With Acute Heart Failure (DAPA-RESPONSE-AHF)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Noha Mansour, Lecturer of Clinical Pharmacy, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-61
Record Dates: First submitted 2021-11-12; First posted 2022-06-06 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Acute Heart Failure
Keywords: Diabetic and non diabetic
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozine 10mg (Experimental)
  Interventions: Drug: Dapagliflozin 10mg Tab
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — patients will receive once daily dapagliflozin 10 mg orally in addition to standard care
  Arms: Dapagliflozine 10mg
Other: Placebo — patients will receive placebo and standard care.
  Arms: Placebo

SUMMARY:
Dapagliflozin, a sodium-glucose cotransporter-2 inhibitor (SGLT2i), increases natriuresis alone and synergistically when combined with loop diuretics in patients with AHF without increasing renin angiotensin- aldosterone activity. Thus, adding SGLT2i to the standard loop diuretic therapy might confer additional decongestive and natriuretic benefits while avoiding the adverse electrolyte abnormalities and neurohormonal activation associated with other diuretic combination. These potential benefits may help with improved clinical outcomes, but clinical evidence is still lacking.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older who are hospitalized for hypervolemic AHF, with evidence of congestion defined as either:

   * 2 of the following signs or symptoms: peripheral edema, ascites, jugular venous pressure > 10mmHg, orthopnea, paroxysmal nocturnal dyspnea, 5-pound weight gain, or signs of congestion on chest x-ray or lung ultrasound.

   OR

   *If pulmonary artery catheterization is available, a pulmonary capillary wedge pressure greater than 19 mmHg plus a systemic physical exam finding of hypervolemia from the list above.
2. Randomized within 24 hours of hospitalization for AHF
3. Planned use of IV loop diuretic therapy during current hospitalization
4. Estimated glomerular filtration rate (eGFR) of at least 30 ml/min/1.73m2 by the MDRD equation
5. For diabetic patients, history of type 2 diabetes or a new hemoglobin A1c 6.5% on admission.

Exclusion Criteria:

1. Type 1 diabetes mellitus.
2. Dyspnea primarily due to non-cardiac causes.
3. Cardiogenic shock.
4. Acute coronary syndrome within 30 days prior to randomization.
5. Planned or recent percutaneous or surgical coronary intervention within 30 days prior to randomization.
6. Signs of ketoacidosis and/or hyperosmolar hyperglycemic syndrome (pH>7.30 and glucose >15 mmol/L and HCO3>18 mmol/L).
7. Pregnant or nursing (lactating) women.
8. Heart failure due to drug toxicity
9. Adherence to medication less than 95%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Change in dyspnea ( Visual analogue scale) (VAS) | From baseline to day 4
  • Comparing the area under the curve (AUC) of change in VAS dyspnea score. To do so, individual changes in VAS score will be visualized as a curve where the x-axis shows study day baseline to day 5, and y-axis shows VAS score. the overall VAS AUC score (mm × h) will be compared across treatment groups

SECONDARY OUTCOMES:
Incidence of worsening heart failure (HF) | From the date of randomization until discharge or end of treatment, whichever came first, assessed up to 30 days
  Defined as worsening signs and/or symptoms of HF that require IV inotropic therapy or admission to an intensive care unit or mechanical ventilatory, renal or circulatory support.
All-cause death | 30 days from discharge
  Difference in all cause mortality rate
All-cause death | 60 days from discharge
  Difference in all cause mortality rate
Hospital readmission | 30 days from discharge
  Difference between groups in rate of readmission after discharge for heart failure related reason
Hospital readmission | 60 days from discharge
  Difference between groups in rate of readmission after discharge for heart failure reason
Urinary sodium 2 hours post randomization | 2 Hours
  Difference in sodium execrated in urine (mmol/L) after 2 hours between study groups
Difference in serum levels of congestion biomarkers | 4 days post-randomization
  Difference in serum levels of Nt-ProBNP 4 days post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Noha Mansour, PhD, Principal Investigator — Department of Clinical Pharmacy & Pharmacy Practice, Faculty of Pharmacy, University of Mansoura; Moheb Magdy Mouris, MD, Principal Investigator — Department of Cardiology, Faculty of Medicine, University of Mansoura; Mohamed El-Husseiny Shams, Proffesor, Study Chair — Department of Clinical Pharmacy & Pharmacy Practice, Faculty of Pharmacy, University of Mansoura
Locations (1):
- Noha Mansour, Al Mansurah, Egypt

REFERENCES:
- [Derived] Emara AN, Wadie M, Mansour NO, Shams MEE. The clinical outcomes of dapagliflozin in patients with acute heart failure: A randomized controlled trial (DAPA-RESPONSE-AHF). Eur J Pharmacol. 2023 Dec 15;961:176179. doi: 10.1016/j.ejphar.2023.176179. Epub 2023 Nov 2. PMID 37923161